CLINICAL TRIAL: NCT02308995
Title: Barbed Sutures Versus Conventional Sutures in Laparoscopic Excision of Endometrioma . A Randomized Controlled Study
Brief Title: Barbed Sutures Versus Conventional Sutures in Laparoscopic Excision of Endometrioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Prof .Usama M.Fouda, M.D, PhD, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lap.cystectomy.barbed
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Laparoscopy; Barbed sutures
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cystectomy using barbed sutures (Experimental): Endometrioma bed is sutured with barbed sutures
  Interventions: Procedure: Cystectomy using barbed sutures; Device: V-Loc (Covidien, Mansfield, MA)
- Cystectomy using conventional sutures (Active Comparator): Endometrioma bed is sutured with conventional sutures
  Interventions: Procedure: Cystectomy using conventional sutures; Device: polyglactin 910 suture(VICRYL™, Ethicon Inc, Sommerville, NJ)

INTERVENTIONS:
Procedure: Cystectomy using barbed sutures — A sharp transverse cortical incision was made over the endometroma using unipolar hook and a cleavage plane was developed by sharp dissection. After the identification of the cleavage plane, the entire cyst will be enucleated by means of adequate traction with a strong grasper and counter-traction maneuvers with another grasping forceps . The ovarian edges will be re-approximated by using V-Loc (Covidien, Mansfield, MA).
  Arms: Cystectomy using barbed sutures
Procedure: Cystectomy using conventional sutures — A sharp transverse cortical incision was made over the endometroma using unipolar hook and a cleavage plane was developed by sharp dissection. After the identification of the cleavage plane, the entire cyst will be enucleated by means of adequate traction with a strong grasper and counter-traction maneuvers with another grasping forceps . The ovarian edges will be re-approximated by using polyglactin 910 suture(VICRYL™.; Ethicon Inc, Sommerville, NJ) .
  Arms: Cystectomy using conventional sutures
Device: V-Loc (Covidien, Mansfield, MA)
  Arms: Cystectomy using barbed sutures
Device: polyglactin 910 suture(VICRYL™, Ethicon Inc, Sommerville, NJ)
  Arms: Cystectomy using conventional sutures

SUMMARY:
The aim of this randomized controlled trial is to compare operative data and early postoperative outcomes of laparoscopic excision of endometrioma using barbed sutures with those of laparoscopic excision of endometrioma using conventional sutures.

DETAILED DESCRIPTION:
Several authors reported the use of barbed sutures in myomectomy , hysterectomy and closure of vaginal vault. A recent meta-analysis comparing the efficacy of laparoscopic suturing using barbed suture or conventional sutures in myomectomy or hysterectomy revealed that suturing with barbed sutures was associated with less suturing time and operative time.

Although numerous studies revealed the advantages of using barbed sutures , no studies have yet evaluated the use of barbed sutures in laparoscopic excision of endometrioma.

The aim of this randomized controlled trial is to compare operative data and early postoperative outcomes of laparoscopic excision of endometrioma using barbed sutures with those of laparoscopic excision of endometrioma using conventional sutures.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral endometrioma more than 3 cm in mean diameter

Exclusion Criteria:

* Bilateral endometriomata
* Conversion of laparoscopy to laparotomy
* Contraindications for general anesthesia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Suturing time of endometrioma bed | During cystectomy operation

SECONDARY OUTCOMES:
Operative time | During cystectomy operation

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Aljazeera Hospital
Locations (1):
- Aljazeera hospital, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided